CLINICAL TRIAL: NCT02326974
Title: The Impact of HER2 Heterogeneity on the Treatment of Early-stage HER2-positive Breast Cancer: a Phase II Study of T-DM1 in Combination With Pertuzumab in the Preoperative Setting
Brief Title: T-DM1+Pertuzumab in Pre-OP Early-Stage HER2+ BRCA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Otto Metzger, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-409
Record Dates: First submitted 2014-12-15; First posted 2014-12-30 (Estimated); Results first posted 2021-05-11 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: HER-2 Positive Breast Cancer; Breast Cancer; Stage II Breast Cancer; Stage III Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine; pertuzumab; Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- T-DM1 and Pertuzumab (Experimental): T-DM1 3.6 mg per kg of body weight via IV every 3 weeks for 6 doses and Pertuzumab loading dose of 840 mg via IV on Cycle 1 Day 1 followed by maintenance dose of 420 mg via IV every 3 weeks for 6 doses. Excision of tumor/mastectomy of biopsy residual tumor within 42 days of the last cycle of therapy.
  Interventions: Drug: T-DM1; Drug: Pertuzumab; Procedure: Excision of tumor/mastectomy

INTERVENTIONS:
Drug: T-DM1 — Neoadjuvant treatment is for a total of 18 weeks.
  Other Names: Kadcyla
Drug: Pertuzumab — Neoadjuvant treatment is for a total of 18 weeks.
  Other Names: Perjeta
Procedure: Excision of tumor/mastectomy — Definitive breast cancer surgery (excision or mastectomy) marks the end of protocol mandated therapy.

SUMMARY:
This research study is studying a combination of drugs as a possible treatment for breast cancer that has tested positive for a protein called HER2.

The names of the study interventions involved in this study are:

* Trastuzumab emtansine (also called T-DM1)
* Pertuzumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied. The FDA (the U.S. Food and Drug Administration) has not approved T-DM1 for pre-operative use in breast cancer but it has been approved for other uses in breast cancer. The FDA has approved pertuzumab as a pre-operative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have HER2-positive Stage II or III histologically confirmed invasive carcinoma of the breast. A minimum tumor size of 2 cm determined by physical exam or imaging is required.
* HER-2 positive, confirmed by central testing (Clarient labs): IHC 3+ and/or FISH positive based on one of the three following criteria:
* Single-probe average HER2 copy number≥6.0 signals/cell OR
* Dual-probe HER2/CEP17 <2.0 with an average HER2 copy number ≥6.0 signals/cell OR
* Dual-probe HER2/CEP17 ratio ≥2.0
* ER/PR determination is required.
* Bilateral breast cancers are allowed if both cancers are HER2-positive.
* Patients with multifocal or multicentric disease are eligible as long as one area meets eligibility criteria.
* Breast imaging should include the ipsilateral axilla. For subjects with a clinically negative axilla, a sentinel lymph node biopsy will be performed either before or after preoperative therapy at the discretion of the subject's physicians. For subjects with a clinically positive axilla, a needle aspiration, core biopsy or SLN procedure will be performed to determine the presence of metastatic disease in the lymph nodes.
* Men and women (with any menopausal status) ≥ 18 years of age
* ECOG performance status 0 or 1
* Required laboratory values:

  * ANC ≥1500/mm3
  * Hemoglobin ≥ 9 g/dl
  * Platelets ≥100,000/mm3
  * Serum creatinine < 1.5 X ULN (institutional)
  * Total bilirubin ≤ 1.0 X ULN (institutional) For patients with Gilbert syndrome, the direct bilirubin should be within the institutional normal range.
  * AST and ALT ≤ 1.5x ULN (institutional)
  * Alkaline phosphatase ≤1.5x ULN (institutional)
* Documentation of hepatitis B virus (HBV) and hepatitis C virus (HCV) serologies is required: this includes hepatitis B surface antigen (HBsAg) and/or total hepatitis B core antibody (HBcAb) in addition to HCV antibody testing.
* Only for patients who test positive for hep B/C virus: PTT/INR < ULN (institutional)
* Left ventricular ejection fraction (LVEF) ≥ 55%
* Premenopausal women must have a negative serum pregnancy test, including women who have had a tubal ligation and for women less than 12 months after the onset of menopause.
* Women of childbearing potential and men with partners of childbearing potential must be willing to use one highly effective form of non-hormonal contraception or two effective forms of non-hormonal contraception by the patient and/or partner and continue its use for the duration of the study treatment and for 7 months after the last dose of study treatment.
* Potent CYP3A4 inhibitors, such as ketoconazole and erythromycin, should be avoided during the study treatment period with T-DM1.
* Excessive alcohol intake should be avoided (occasional use is permitted).
* Patients with a history of ipsilateral DCIS are eligible.
* Patients undergoing breast conservation therapy (i.e. lumpectomy) must not have any contraindications to radiation therapy.
* Willing and able to sign informed consent.
* Willing to provide tissue for research purposes.

Exclusion Criteria:

* Pregnant or nursing women due to the teratogenic potential of the study drugs.
* Active, unresolved infection.
* Receipt of intravenous antibiotics for infection within 7 days prior to enrollment.
* Patients with active liver disease, for example, due to hepatitis B virus, hepatitis C virus, autoimmune hepatic disorder, or sclerosing cholangitis.
* Uncontrolled hypertension (systolic >180 mm Hg and/or diastolic >100 mm Hg) or clinically significant (i.e. active) cardiovascular disease: cerebrovascular accident/stroke or myocardial infarction within 6 months prior to first study medication, unstable angina, congestive heart failure (CHF) of New York Heart Association (NYHA) Grade II or higher, or serious cardiac arrhythmia requiring medication.
* Significant symptoms (Grade ≥2) peripheral neuropathy.
* Other concurrent serious diseases that may interfere with planned treatment, including severe pulmonary conditions/illness, uncontrolled infections, uncontrolled diabetes.
* Any prior treatment for the current breast cancer, including chemotherapy, hormonal therapy, radiation or experimental therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2028-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Otto Metzger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Tennessee Oncology/Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- [Derived] Li Z, Metzger Filho O, Viale G, dell'Orto P, Russo L, Goyette MA, Kamat A, Yardley DA, Gupta Abramson V, Arteaga CL, Spring LM, Chiotti K, Halsey C, Waks AG, King TA, Lester SC, Bellon JR, Winer EP, Spellman PT, Krop IE, Polyak K. HER2 heterogeneity and treatment response-associated profiles in HER2-positive breast cancer in the NCT02326974 clinical trial. J Clin Invest. 2024 Feb 1;134(7):e176454. doi: 10.1172/JCI176454. PMID 38300710

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from January 2015 to January 2018.
Period: Overall Study
Arm/Group | T-DM1 and Pertuzumab
Started | 164
Treated | 163
Completed | 157
Not Completed | 7
Not completed — Withdrawal by Subject | 2
Not completed — failed heterogenity evaluation | 5

BASELINE CHARACTERISTICS:
Population: patients treated with at least one dose of T-DM1 and pertuzumab
Arm/Group | T-DM1 and Pertuzumab
Number analyzed (Participants) | 163
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 131
  >=65 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 147
  Unknown or Not Reported | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 139
  More than one race | 1
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 163
Hormone Receptor Status [Count of Participants; unit: Participants] — Estrogen Receptor (ER) and Progesterone Receptor (PR) status
  Participants
    ER+ and/or PR+ | 112
    ER- and PR- | 41
HER2 Amplification Status [Count of Participants; unit: Participants] — Patients underwent two ultrasound-guided core biopsies from different geographic areas of the same tumor prior to treatment. Central pathology evaluation of intratumor heterogeneity of HER2 expression was assessed by fluorescence in situ hybridization (FISH). HER2 heterogeneity was defined following the College of American Pathologists and the United Kingdom guidelines. HER2 heterogeneity was defined as the existence of an area of tumor cells with HER2 amplification representing more than 5% but less than 50% of infiltrating tumor cells, or an area of tumor that tested HER2-negative by FISH.
  Participants
    Heterogenous | 16
    Non-Heterogenous | 141
    Missing | 6
Clinical Stage [Count of Participants; unit: Participants] — Defined as the clinical breast cancer stage at baseline. Stage is degree of cancer burden, including size of cancer and nodal involvement. Stage 1 is the least burden and stage 2 and 3 having increased burden.
  Participants
    Stage 1 | 1
    Stage 2 | 138
    Stage 3 | 24
HER-2 results by IHC (central confirmation) [Count of Participants; unit: Participants] — HER-2 results by IHC confirmed by central laboratory. HER-2 status by immunohistochemistry with 3+ indicating clear HER-2 protein overexpression and 2+ indicating an equivocal level of HER-2 expression.
  HER2: human epidermal growth factor receptor 2
  Participants
    2+ | 40
    3+ | 121
    Unknown | 2
Histologic Grade [Count of Participants; unit: Participants] — Histologic grade is a measure of cancer differentiation. Grade 1 is well differentiated, grade 2 is moderate differentiated and grade 3 is poorly differentiated.
  Participants
    Grade 1 | 3
    Grade 2 | 56
    Grade 3 | 103
    Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Pathologic Complete Response (pCR) by HER2 Amplification Status Non-Heterogeneous
Description: The rate of pCR is the percentage of participants with Residual Cancer Burden (RCB)=0 as defined by established guidelines (Symmans et al. JCO 2007; M.D Anderson http://www.mdanderson.org/breastcancer_RCB).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Evaluate upon completion of breast surgery, up to approximately 24 weeks from study enrollment.
Population: Patients treated with at least one dose of T-DM1 and Pertuzumab and evaluable (with invasive disease present on the research core biopsy for evaluation of HER-2 heterogeneity by central pathology evaluation).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Heterogeneous HER2 Amplification Status: T-DM1 and Pertuzumab T-DM1 3.6 mg per kg of body weight via IV every 3 weeks for 6 doses and Pertuzumab loading dose of 840 mg via IV on Cycle 1 Day 1 followed by maintenance dose of 420 mg via IV every 3 weeks for 6 doses. Excision of tumor/mastectomy of biopsy residual tumor within 42 days of the last cycle of therapy.
- Non-Heterogeneous HER2 Amplification Status: T-DM1 3.6 mg per kg of body weight via IV every 3 weeks for 6 doses and Pertuzumab loading dose of 840 mg via IV on Cycle 1 Day 1 followed by maintenance dose of 420 mg via IV every 3 weeks for 6 doses. Excision of tumor/mastectomy of biopsy residual tumor within 42 days of the last cycle of therapy.
Arm/Group | Heterogeneous HER2 Amplification Status | Non-Heterogeneous HER2 Amplification Status
Number analyzed (Participants) | 16 | 141
percentage of participants | 0 [0 to 20.6] | 54.6 [46.0 to 63.0]
Statistical Analysis 1: Comparison: Heterogeneous HER2 Amplification Status vs Non-Heterogeneous HER2 Amplification Status; By estimating that the overall pCR with T-DM1 plus pertuzumab would be approximately 40%, and 20% of the population classified as heterogeneous, the study would have 80% power with 136 evaluable patients to detect a difference in pCR of 44.9% in the non-heterogenous versus 20.3% in the heterogenous subgroup. The study had a 90% power to detect difference in pCR of 43.4% in the non-heterogenous versus 8.8% in the heterogenous subgroup if the observed prevalence of HER2 heterogeneity was 10%; Test type: Superiority; p < 0.001, Mantel Haenszel

2. Secondary Outcome: Rate of Pathologic Complete Response (pCR)
Description: The rate of pCR is the percentage of participants with Residual Cancer Burden (RCB)=0 as defined by established guidelines (Symmans et al. JCO 2007; M.D Anderson http://www.mdanderson.org/breastcancer_RCB).
Time Frame: Evaluate upon completion of breast surgery, up to approximately 24 weeks from study enrollment.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T-DM1 and Pertuzumab
Number analyzed (Participants) | 157
percentage of participants | 49.0 [41.0 to 57.1]

3. Secondary Outcome: Hormone Receptor (HR) Status by HER2 Amplification Status
Description: HR status classified by estrogen receptor (ER) and/or progesterone receptor (ER) positive versus ER negative and PR negative determined by immunohistochemical methods according to the local institution's standard protocol.
Time Frame: Day 0 (baseline/at study entry)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Non-Heterogeneous HER2 Amplification Status: T-DM1 and Pertuzumab T-DM1 3.6 mg per kg of body weight via IV every 3 weeks for 6 doses and Pertuzumab loading dose of 840 mg via IV on Cycle 1 Day 1 followed by maintenance dose of 420 mg via IV every 3 weeks for 6 doses. Excision of tumor/mastectomy of biopsy residual tumor within 42 days of the last cycle of therapy.
Arm/Group | Heterogeneous HER2 Amplification Status | Non-Heterogeneous HER2 Amplification Status
Number analyzed (Participants) | 16 | 141
Participants
  HR-positive | 13 | 96
  HR-negative | 3 | 45

4. Secondary Outcome: Median Disease-Free Survival
Description: Disease-free survival (DFS) based on the Kaplan-Meier method is defined as the duration of time from study entry to the occurrence of the first of the following events: local/regional recurrence, contralateral invasive breast cancer, distant recurrence or death from any cause. In situ cancer is not included as DFS event. Participants alive without an event are censored at date of last disease assessment.
Time Frame: Post-surgery follow-up of disease and survival occurs every 6 months for 5 years and annually until year 10.
Reporting Status: Not Posted, anticipated posting 2028-01

5. Secondary Outcome: Median Overall Survival
Description: Overall survival (OS) based on Kaplan-Meier methods is defined as the interval from the date of registration to death from any cause. Patients are censored at date last known alive.
Time Frame: Post-surgery follow-up of disease and survival occurs every 6 months for 5 years and annually until year 10.
Reporting Status: Not Posted, anticipated posting 2028-01

6. Secondary Outcome: Clinical Response Rate (Complete Response)
Description: Clinical response rate was defined as the percentage of participants achieving complete response (CR) based on RECIST 1.1 criteria on treatment up to surgery. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions
Time Frame: Evaluate upon completion of neoadjuvant therapy, up to approximately 18 weeks from study enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | T-DM1 and Pertuzumab
Number analyzed (Participants) | 163
Participants | 62

7. Secondary Outcome: Clinical Response Rate (Partial Response)
Description: Clinical response rate was defined as the percentage of participants achieving partial response (PR) based on RECIST 1.1 criteria on treatment up to surgery. Per RECIST 1.1 for target lesions: PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD.
Time Frame: Evaluate upon completion of neoadjuvant therapy, up to approximately 18 weeks from study enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | T-DM1 and Pertuzumab
Number analyzed (Participants) | 163
Participants | 69

8. Secondary Outcome: Number of Participants With a Dose Reduction
Description: Number of participants with ever having dose reduction on neoadjuvant therapy up to surgery.
Time Frame: Evaluate upon completion of neoadjuvant therapy, up to approximately 18 weeks from study enrollment.
Population: Patients treated with at least one dose of T-DM1 and Pertuzumab.
Measure: Count of Participants; unit: Participants
Arm/Group | T-DM1 and Pertuzumab
Number analyzed (Participants) | 163
Participants | 18

9. Secondary Outcome: Treatment-Emergent Fatigue Rate
Description: Treatment-emergent fatigue rate is the percentage of participants who experienced grade 1-2 fatigue based on the Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0 as reported on the adverse event case report form. CTCAE severity scale ranges from 0 (none) to 5 (death): Grade 1=mild and Grade 2=moderate.
Time Frame: Adverse events are assessed every cycle of neoadjuvant therapy prior to surgery, up to approximately 18 weeks (6 cycles) from study enrollment.
Population: Patients treated with at least one dose of T-DM1 and Pertuzumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | T-DM1 and Pertuzumab
Number analyzed (Participants) | 163
percentage of participants | 76.1 [68.8 to 82.4]

ADVERSE EVENTS:
Time Frame: Adverse events are assessed every cycle of neoadjuvant therapy prior to surgery, up to approximately 18 weeks (6 cycles) from study enrollment.
Description: Serious adverse events (AEs) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Maximum grade toxicity by type for a patient over time was calculated. No further data is available to specify classification of other beyond the general term.
Groups:
- T-DM1 and Pertuzumab: T-DM1 via IV every 3 weeks for 6 doses and Pertuzumab loading dose via IV on Cycle 1 Day 1 followed by maintenance dose via IV every 3 weeks for 6 doses. Excision of tumor/mastectomy of biopsy residual tumor
  T-DM1: Participants will receive Trastuzumab emtansine (T-DM1) by IV every 3 weeks for 6 doses; for a total of 18 weeks of treatment.
  Pertuzumab: Participants will receive a loading dose of pertuzumab by IV on Cycle 1 Day 1 followed by maintenance dose of pertuzumab by IV every 3 weeks for a total of 6 doses; for a total of 18 weeks of treatment.
  Excision of tumor/mastectomy: Definitive breast cancer surgery (excision or mastectomy) marks the end of protocol mandated therapy.
Arm/Group | T-DM1 and Pertuzumab
All-Cause Mortality (participants affected / at risk) | 0/163
Serious Adverse Events (participants affected / at risk) | 11/163
Other Adverse Events (participants affected / at risk) | 162/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T-DM1 and Pertuzumab (N=163)
Anemia (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 1
Platelet count decreased (Investigations) | 2
Hypokalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T-DM1 and Pertuzumab (N=163)
Anemia (Blood and lymphatic system disorders) | 27
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2
Mitral valve disease (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 5
Sinus tachycardia (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 3
Middle ear inflammation (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 2
Hypothyroidism (Endocrine disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Chills (General disorders) | 2
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 81
Fever (General disorders) | 3
Flu like symptoms (General disorders) | 4
Infusion related reaction (General disorders) | 3
Non-cardiac chest pain (General disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT02326974/Prot_SAP_000.pdf